CLINICAL TRIAL: NCT02555462
Title: Real-Ear Measurement (REM) and Test Box System Integration Into Fitting Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phonak AG, Switzerland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KEK-ZH-NR.2015-0099
Record Dates: First submitted 2015-09-14; First posted 2015-09-21 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Validation Studies

ARMS (1):
- Real-Ear Measurement (Experimental): The study arm goes through a comparative test run followed by a comparative hearing aid fitting.
  Interventions: Device: Real-Ear Measurement system integrated in hearing aid fitting software

INTERVENTIONS:
Device: Real-Ear Measurement system integrated in hearing aid fitting software — The subjects individual response of the ear canal gets measured with the help of a probe tube and a following hearing aid fitting.

SUMMARY:
Integration of the REM-verification within the fitting workflow will enable the hearing care professional to easily run real ear measurements. The purpose of the two study parts is to prove that an integrated cooperative system, consisting of fitting software and measurement system, matches desired responses for certain stimuli faster, more reliably and more precisely at the ear drums of hearing instrument wearers than current best practice processes.

ELIGIBILITY:
Inclusion Criteria:

* Clean and healthy ear canal, eardrum and pinna
* Ability to keep current position (of head and body) during a period of about 5 minutes while seated.

Exclusion Criteria:

* Ear infections
* Ear wax in the ear
* Hyperacusis
* Pacemaker
* Tremor
* Disability to keep position.

Ages: 16 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Distance (mm) from probe tube to eardrum measurement | 1 month
  Precise of the Probe Tube placement
Procedure time (min) of fitting workflow including Real Ear measurement | 2 month
  In addition to the outcome measurement "time" (in minutes) further outcome measurements can be obtained due to the performed real ear measurement procedure itself.
  Data that give information pertaining to test reliability (in dB) and precision of hearing aid fitting (in dB).

SECONDARY OUTCOMES:
Subjective rating of unpleasantness (0 = not unpleasant at all, 10 = very unpleasant) | 1 month
  Pleasantness during the probe tube placement
Questionnaire about perceived annoyance | 2 month
  Perceived annoyance of the hearing care professional and the test subject measured with a questionnaire including rating scales for stessful and boring.

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak AG, Stäfa, Canton of Zurich, Switzerland